CLINICAL TRIAL: NCT04912427
Title: A Phase Ib Study of Isatuximab, Velcade, and Dexamethasone in Patients With Multiple Myeloma and Severe KIDNEY Disease
Brief Title: Isatuximab, Velcade, and Dexamethasone in Patients With Multiple Myeloma and Severe KIDNEY Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202107134
Record Dates: First submitted 2021-05-27; First posted 2021-06-03 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isatuximab + Boretezomib + Dexamethasone (Experimental): * Each cycle is 28 days
  * Cycle 1
    * Days 1, 8, 15, and 22: Dexamethasone at start time, Bortezomib at 30 minutes after start time, and Isatuximab at 60 minutes after start time
  * Cycles 2-8
    * Days 1 and 15: Dexamethasone at start time, Bortezomib at 30 minutes after start time, and Isatuximab at 60 minutes after start time
    * Days 8 and 22: Dexamethasone at start time and Bortezomib at 30 minutes after start time
  * Cycles 9+
    * Days 1 and 15: Dexamethasone at start time and Isatuximab at 30-60 minutes after start time
  Interventions: Drug: Isatuximab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Isatuximab is supplied by Sanofi.
  Other Names: Sarclisa
Drug: Bortezomib — Bortezomib is commercially available.
  Other Names: Velcade
Drug: Dexamethasone — Dexamethasone is commercially available.

SUMMARY:
This is a phase Ib study to assess the safety, tolerability, preliminary efficacy, and renal response of isatuximab, bortezomib, and dexamethasone in newly diagnosed multiple myeloma patients with severe renal impairment or dialysis-dependent end-stage renal disease. Such patients have limited therapeutic options due to renal clearance or nephrotoxicity of many myeloma therapies and are often excluded from clinical trials. Isatuximab in other regimens has shown efficacy and tolerability in patients with moderate renal impairment, although data are lacking for regimens containing CD38-targeting immunotherapies in severe renal impairment/ESRD.

ELIGIBILITY:
Inclusion Criteria:

This study will enroll 28 evaluable patients. Fourteen (+/- 2) patients will be required tto be on dialysis and 14 (+/- 2) patients will not be on dialysis.

* Newly diagnosed multiple myeloma diagnosis according to IMWG criteria. Patients eligible for autologous stem cell transplant may be enrolled if the intent is to proceed to transplant after 4 or more cycles of study treatment.
* Severe renal impairment (eGFR < 30ml/min/1.73m^2 using the MDRD calculator) or on dialysis. The value at screening confirms eligibility (if eGFR improves prior to enrollment, this does not render a patient ineligible) The renal impairment may be acute or chronic and may be related to the underlying myeloma (e.g. multiple myeloma (MM) cast nephropathy, monoclonal immunoglobulin deposition disease [MIDD], myeloma cell infiltration) or another cause (e.g. diabetes, hypertension), however the acuity/chronicity and the underlying cause should be documented clearly. Those who have acute kidney injury from hypercalcemia should receive intravenous hydration and calcium-lowering therapy to see if this renal impairment is reversible.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mm3 (growth factor to achieve this level is permissible)
  * Platelets ≥ 50,000/mm3 (transfusion to achieve this level is permissible)
  * Bilirubin ≤ 2 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 3.5 x institutional upper limit of normal (IULN)
* The effects of isatuximab and bortezomib on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 5 months after discontinuation of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 5 months after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Concomitant use of other anti-neoplastic medications or radiotherapy (except for localized disease). Note: Participants are permitted to have received one dose of bortezomib or up to 80 mg of dexamethasone (or equivalent) prior to study treatment initiation if deemed clinically necessary for disease control.
* Currently receiving any other investigational agents.
* Evidence of myeloma within the CNS
* Presence of amyloidosis without concomitant multiple myeloma. Patients with concomitant amyloidosis and multiple myeloma are eligible.
* Prior refractoriness, intolerance or hypersensitivity to bortezomib.
* Prior treatment with an anti-CD38 monoclonal antibody.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to isatuximab, bortezomib, or dexamethasone or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Active acute or chronic hepatitis B viral infection.

  * Screening with serological tests for HBV with surface antigen and antibody (HBsAg and HBsAb) and HBV total core antibody (HBcAb IgG and IgM), and screening for HCV (HCV Ab and HCV RNA level) are required to have been performed within 1 year of screening, or should otherwise be performed as part of screening.
  * Patients with uncontrolled or active HBV infection (patients with positive HBsAg and/or HBV DNA), as well as patients with active HCV infection (positive HCV RNA and negative anti-HCV) are not eligible
  * In case HBcAb are positive, HBV DNA testing by polymerase chain reaction will also be done at baseline. For patients with positive anti-HBc IgG, negative HBsAg and undetectable (under limit of quantification) HBV DNA at study entry (HBV carriers: past resolved infection, resolving acute infection or receiving antiviral treatment with controlled infection), specialist advice may be requested, close monitoring of viral reactivation throughout and following the end of study treatment should be proposed (alanine aminotransferase, aspartate aminotransferase, and HBV DNA at least every 3 months, up to 6 months after treatment discontinuation or initiation of further anticancer therapy.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Baseline Grade 2 or higher peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the regimen as measured by the proportion of patients that discontinue therapy before Cycle 3 for toxicity or intolerance | Through completion of cycle 3 for all enrolled patients (estimated to be 39 months)
  -Patients who discontinue therapy due to COVID-19 will not be included in the calculation of this proportion and will be replaced. Patients who discontinue therapy due to progressive disease before initiation of Cycle 3 will be replaced in the trial.

SECONDARY OUTCOMES:
Renal response per IMWG criteria | Through completion of treatment (estimated to be 6 months)
  * Dialysis dependent at enrollment:
    * Conversion to dialysis independence: Return of renal function to where dialysis is not required for at least one consecutive month
    * Sustained dialysis independence: Return of renal function to where dialysis is not required for at least six consecutive months
  * Dialysis -independence at baseline or achieved while on therapy:
    * Complete response: Improved CrCl ≥ 60 mL/min
    * Partial response: In patients with baseline eGFR < 15mL/min/1.73 m2, CrCl improved to 30 to 59 mL/min
    * Minor response: if baseline eGFR < 15mL/min/1.73 m2, CrCl improved to 15 to 29 mL/min or if baseline eGFR 15 - 29 mL/min/1.73 m2, CrCl improved to 30 to 59 mL/min
    * Progressive renal disease: requirement of sustained
Overall response rate (ORR) per IMWG criteria | Through completion of treatment (estimated to be 6 months)
  -Partial response or better includes minimal residual disease (MRD) - negative, stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response per IMWG criteria
Progression-free survival (PFS) | From cycle 1 day 1 through 5 years after completion of treatment (estimated to be 5 years and 6 months)
  * PFS is defined as time from cycle 1 day 1 until progressive disease or death from any cause
  * Progressive disease is defined by IMWG Criteria
Overall survival (OS) | From cycle 1 day 1 through 5 years after completion of treatment (estimated to be 5 years and 6 months)
  -OS is defined as the time from cycle 1 day 1 until death from any cause
Duration of response (DOR) | Through completion of treatment (estimated to be 6 months)
  -DOR: for patients who achieve partial response or better, time from response was first noted until time of progressive disease; deaths due to causes other than progression are censored.
Safety and tolerability of regimen as measured by discontinuation rate of each individual drug and duration/dose level exposure for each drug | Through completion of treatment (estimated to be 6 months)
Total number of adverse events | From start of treatment through 30 days after last day of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Total number of treatment-emergent adverse events | From start of treatment through 30 days after last day of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Total number of grade 3 or higher adverse events | From start of treatment through 30 days after last day of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Change in quality of life as measured by the EORTC-QLQ 30 questionnaire | Baseline, end of cycle 1 (each cycle is 28 days), and end of cycle 3 (each cycle is 28 days)
  The EORTC QLQ-C30 comprises 6 functional scales (role function, physical functioning, cognitive functioning, emotional functioning, social functioning and global quality of life) as well as nine symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). With the exception of 2 items included in the global health/quality of life scale, for which responses range from 1 (Very poor) to 7 (Excellent), item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores for all functional scales and Global Health Status indicate better quality of life; increase from baseline indicates improvement in quality of life compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stockerl-Goldstein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu